CLINICAL TRIAL: NCT00263380
Title: Experimental Study on the Role of Corticosteroids and Beta-Agonists on Cytokine Production in COPD Patients
Brief Title: Investigation on the Role of Corticosteroids and Beta-Agonists on Cytokine Production in COPD Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Antonius Hospital (Other)
Other Study IDs: COPD IL8
Record Dates: First submitted 2005-12-07; First posted 2005-12-08 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2005-07

CONDITIONS: COPD
Keywords: COPD; cytokines; corticosteroids; beta agonists; synergistic effect
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Research on the synergistic effect of corticosteroids and beta-agonists on the cytokine production in COPD patients. Blood will be obtained from healthy volunteers and COPD patients and blood monocytes will be stimulated to produce cytokines with or without the prementioned drugs.

ELIGIBILITY:
Inclusion Criteria:

* clinical COPD
* smoking
* age > 40 years

Exclusion Criteria:

* age < 40 years
* use of antibiotics, corticosteroids or beta-agonists

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2005-10

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ten Broeke, Dr, Principal Investigator — St. Antonius Hospital
Locations (1):
- St Antonius Hospital, Nieuwegein, Utrecht, Netherlands